CLINICAL TRIAL: NCT05938920
Title: A Phase IIa, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Efficacy of INS018_055 Administered Orally to Subjects With Idiopathic Pulmonary Fibrosis (IPF)
Brief Title: Study Evaluating INS018_055 Administered Orally to Subjects With Idiopathic Pulmonary Fibrosis (IPF)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: InSilico Medicine Hong Kong Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INS018-055-003
Record Dates: First submitted 2023-06-28; First posted 2023-07-11 (Actual); Results first posted 2025-12-02 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Idiopathic Pulmonary Fibrosis (IPF)
Keywords: Pulmonary Fibrosis; Idiopathic Pulmonary Fibrosis; Fibrosis; Pathologic Processes; Lung Diseases, Interstitial; Lung Diseases; Respiratory Tract Diseases
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Pulmonary Fibrosis; Fibrosis; Pathologic Processes; Lung Diseases, Interstitial; Lung Diseases; Respiratory Tract Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- INS018_055 30 mg QD (Experimental): Group 1: INS018_055 once daily up to 12 weeks, low dose
  Interventions: Drug: INS018_055
- INS018_055 30 mg BID (Experimental): Group 2: INS018_055 twice daily up to 12 weeks, low dose
  Interventions: Drug: INS018_055
- INS018_055 60 mg QD (Experimental): Group 3: INS018_055 once daily up to 12 weeks, high dose
  Interventions: Drug: INS018_055
- Placebo (Placebo Comparator): Group 4: Placebo once or twice daily up to 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: INS018_055 — Pharmaceutical formulation: Capsules
  Mode of Administration: Oral
  Arms: INS018_055 30 mg BID; INS018_055 30 mg QD; INS018_055 60 mg QD
Drug: Placebo — Pharmaceutical formulation: Capsules
  Mode of Administration: Oral
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn about INS018_055 in adults with Idiopathic Pulmonary Fibrosis (IPF).

The primary objective is to evaluate the safety and tolerability of INS018_055 orally administered for up to 12 weeks in adult subjects with IPF compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged ≥40 years based on the date of the written informed consent form
2. Diagnosis of IPF as defined by American Thoracic Society/European Respiratory Society/Japanese Respiratory Society/Latin American Thoracic Association guidelines
3. In a stable condition and suitable for study participation based on the results of medical history, physical examination, vital signs, 12-lead ECG, and laboratory evaluation
4. Subjects with background pirfenidone or nintedanib may be enrolled if their regimen of antifibrotic therapy has been stable for > 8 weeks prior to Visit 1
5. Meeting all of the following criteria during the screening period:

   1. FVC ≥40% predicted of normal
   2. DLCO corrected for Hgb ≥25% and <80% predicted of normal.
   3. forced expiratory volume in the first second/FVC (FEV1/FVC) ratio >0.7 based on pre-bronchodilator value

Exclusion Criteria:

1. Acute IPF exacerbation within 4 months prior to Visit 1 and/or during the screening period, as determined by the investigator
2. Patients who are unwilling to refrain from smoking within 3 months prior to screening and until the end of the study
3. Female patients who are pregnant or nursing
4. Abnormal ECG findings

Other protocol inclusion and exclusion criteria may apply.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2023-06-19 (Actual); Primary Completion 2024-08-08 (Actual); Study Completion 2024-08-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (22):
- China (22):
  - Anhui Chest Hospital, Hefei, Anhui
  - The Second Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Peking University Shougang Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Hainan General Hospital, Haikou, Hainan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - The Shengjing Hospital of China medical university, Shenyang, Liaoning
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Zhongshan hospital Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - The West China Hospital of Sichuan University, Chengdu, Sichuan
  - General Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital - Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xu Z, Ren F, Wang P, Cao J, Tan C, Ma D, Zhao L, Dai J, Ding Y, Fang H, Li H, Liu H, Luo F, Meng Y, Pan P, Xiang P, Xiao Z, Rao S, Satler C, Liu S, Lv Y, Zhao H, Chen S, Cui H, Korzinkin M, Gennert D, Zhavoronkov A. A generative AI-discovered TNIK inhibitor for idiopathic pulmonary fibrosis: a randomized phase 2a trial. Nat Med. 2025 Aug;31(8):2602-2610. doi: 10.1038/s41591-025-03743-2. Epub 2025 Jun 3. PMID 40461817

RESULTS

PARTICIPANT FLOW:
Groups:
- INS018_055 30 mg QD: Group 1: INS018_055 once daily up to 12 weeks, low dose INS018_055: Pharmaceutical formulation: Capsules Mode of administration: Oral
- INS018_055 30 mg BID: Group 2: INS018_055 twice daily up to 12 weeks, low dose INS018_055: Pharmaceutical formulation: Capsules Mode of administration: Oral
- INS018_055 60 mg QD: Group 3: INS018_055 once daily up to 12 weeks, high dose INS018_055: Pharmaceutical formulation: Capsules Mode of administration: Oral
- Placebo: Group 4: Placebo once or twice daily up to 12 weeks INS018_055: Pharmaceutical formulation: Capsules Mode of administration: Oral
Period: Overall Study
Arm/Group | INS018_055 30 mg QD | INS018_055 30 mg BID | INS018_055 60 mg QD | Placebo
Started | 18 | 18 | 18 | 17
Completed | 16 | 14 | 13 | 16
Not Completed | 2 | 4 | 5 | 1
Not completed — Adverse Event | 1 | 3 | 2 | 1
Not completed — Death | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Not completed — Participant Asked to Withdraw from the Trial | 1 | 0 | 0 | 0
Not completed — Participant Withdrew from Treatment and Refused to do Visit 7 Follow Up Visit | 0 | 0 | 1 | 0
Not completed — Participant Refused to Come In | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) Population
Groups:
- Total: Total of all reporting groups
Arm/Group | INS018_055 30 mg QD | INS018_055 30 mg BID | INS018_055 60 mg QD | Placebo | Total
Number analyzed (Participants) | 18 | 18 | 18 | 17 | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.8 (6.99) | 67.2 (7.77) | 65.7 (6.82) | 68.3 (5.28) | 66.7 (6.73)
Age, Customized [Count of Participants; unit: Participants]
  ≤ 65 years | 9 | 7 | 7 | 4 | 27
  > 65 to ≤ 75 years | 7 | 9 | 10 | 13 | 39
  >75 years | 2 | 2 | 1 | 0 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 2 | 2 | 7
  Male | 18 | 15 | 16 | 15 | 64
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 18 | 18 | 18 | 17 | 71
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 18 | 18 | 18 | 17 | 71
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Height at Baseline [Mean (Standard Deviation); unit: centimeters (cm)] | 167.77 (5.549) | 165.78 (7.869) | 166.29 (6.470) | 164.50 (7.874) | 166.11 (6.944)
Weight at Baseline [Mean (Standard Deviation); unit: kilograms (kg)] | 72.27 (7.395) | 67.36 (12.141) | 73.32 (13.547) | 67.69 (12.117) | 70.20 (11.593)
Body Mass Index at Baseline [Mean (Standard Deviation); unit: kg/m2] | 25.66 (2.080) | 24.41 (3.399) | 26.41 (4.128) | 24.96 (3.733) | 25.36 (3.429)
Forced vital capacity (FVC) at Baseline [Mean (Standard Deviation); unit: liters (L)] — Decline (change) in FVC was assessed from Week 0 to Week 12. FVC was assessed using standardized spirometry equipment.
  liters (L) | 2.6961 (0.44422) | 2.6170 (0.66740) | 2.7616 (0.68415) | 2.2456 (0.47359) | 2.5848 (0.60040)
Diffusion capacity of the lung for carbon monoxide (DLCO) (actual) at Baseline [Mean (Standard Deviation); unit: mmol/min/kPa] — DLCO was assessed during the single breath diffusion test. Each study site used its own equipment and conducted all measurements using the same equipment. Baseline measurement (Visit 2) was the reference visit and change in DLCO (actual) from Week 0/Visit 2 to Week 12 was assessed. No more than 3 DLCO sessions were performed during the screening period.
  mmol/min/kPa | 3.7832 (1.03476) | 3.4291 (0.93188) | 3.7561 (1.25320) | 3.6085 (1.08683) | 3.6447 (1.06898)
Diffusion capacity of the lung for carbon monoxide (DLCO) (% predicted) at Baseline [Mean (Standard Deviation); unit: percentage] — DLCO (% predicted) is the percentage of the DLCO that is predicted based on the participant's hemoglobin level. DLCO was assessed during the single breath diffusion test. Each study site used its own equipment and conducted all measurements using the same equipment. Baseline measurement (Visit 2) was the reference visit and change in DLCO% predicted from Week 0/Visit 2 to Week 12 was assessed. No more than 3 DLCO sessions were performed during the screening period.
  percentage | 47.6952 (12.41070) | 45.1767 (10.55849) | 48.9831 (16.53697) | 49.1347 (15.72199) | 47.7279 (13.78235)
6-minute walk distance (6-MWD) test (in meters) at Baseline [Mean (Standard Deviation); unit: meters (m)] — Participants had to rest for 30 minutes prior to performing the 6-minute walk test. The participant was instructed to walk on a flat, hard surface. The walk for 6 minutes was timed. After 6 minutes the distance the participant had walked was measured. Participants graded their level of dyspnea on a scale of 0 (no dyspnea) to 10 (maximal dyspnea) before walking. After walking, they were reminded of the level they selected pre-walk and then asked to grade again their level of dyspnea. Change in 6-MWD in meters, from Week 0 to Week 12 was assessed.
  meters (m) | 420.81 (122.020) | 387.26 (80.066) | 378.04 (76.252) | 393.21 (73.022) | 394.85 (89.806)
Leicester Cough Questionnaire (LCQ) total score at Baseline [Mean (Standard Deviation); unit: scores on a scale] — The LCQ is a 19-item self-administered questionnaire that assesses cough-related quality of life (QoL). Change in LCQ from Week 0 to Weeks 4, 8, and 12 was assessed. It examines 3 domains: physical, psychological, and social. The range for the total score on the LCQ is 3 to 21, and each domain score ranges from 1 to 7. The overall score for the LCQ for each participant was calculated by adding the individual domain scores. A higher score indicates a better QoL.
  scores on a scale | 17.1290 (3.08860) | 16.1677 (3.51858) | 15.7431 (3.70099) | 16.4370 (3.05011) | 16.3682 (3.32222)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Had at Least 1 Treatment-emergent Adverse Event (TEAE)
Description: TEAEs were either events with start date on or after the start of the Treatment Period and up to 17 days after EOT (end of treatment), or events with start date prior to the start of the Treatment Period whose severity worsened on or after the start of the Treatment Period and up to 17 days after EOT.
  CTCAE=Common Terminology Criteria for Adverse Events
Time Frame: From first dose of study drug until end of study (EOS) visit i.e. up to 13 weeks (+10 days)
Population: Safety Population: The safety population included all participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Group 4: Placebo once or twice daily up to 12 weeks
  Placebo: Pharmaceutical formulation: Capsules
  Mode of Administration: Oral
Arm/Group | INS018_055 30 mg QD | INS018_055 30 mg BID | INS018_055 60 mg QD | Placebo
Number analyzed (Participants) | 18 | 18 | 18 | 17
Participants
  Any TEAE | 13 | 15 | 15 | 12
  TEAE with CTCAE grade ≥3 | 3 | 7 | 8 | 4
  TEAE Leading to discontinuation of treatment | 1 | 5 | 4 | 2
  TEAE Leading to death | 0 | 1 | 0 | 0

2. Secondary Outcome: Relative Change From Baseline in Forced Vital Capacity (FVC)
Description: Decline (change) in FVC is presented from Week 0 to Week 12. FVC was assessed using standardized spirometry equipment.
Time Frame: Week 0/Visit 2 up to Week 12
Population: Intent-to-treat Population: The ITT population included any randomized participant. The ITT Population was used for summary of demographic and baseline characteristics, and it was used for analysis of secondary endpoints except PK analysis
Measure: Mean (Standard Deviation); unit: percentage change in FVC
Arm/Group | INS018_055 30 mg QD | INS018_055 30 mg BID | INS018_055 60 mg QD | Placebo
Number analyzed (Participants) | 13 | 12 | 10 | 14
percentage change in FVC | -0.7923 (3.90508) | 0.6821 (6.09585) | 3.2253 (5.27457) | -0.7126 (8.17452)
Statistical Analysis 1: Comparison: INS018_055 30 mg QD; Test type: Other; Least Squares Mean = -0.6098, 95% CI 2-sided [-4.1026 to 2.8831], Standard Error of Mean 1.78193
Statistical Analysis 2: Comparison: INS018_055 30 mg BID; Test type: Other; Least Squares Mean = 0.6721, 95% CI 2-sided [-3.0738 to 4.4179], Standard Error of Mean 1.91075
Statistical Analysis 3: Comparison: INS018_055 60 mg QD; Test type: Other; Least Squares Mean = 2.8232, 95% CI 2-sided [-1.6970 to 7.3433], Standard Error of Mean 2.30479
Statistical Analysis 4: Comparison: Placebo; Test type: Other; Least Squares Mean = -0.2933, 95% CI 2-sided [-4.5273 to 3.9408], Standard Error of Mean 2.15954

3. Secondary Outcome: Absolute Change From Baseline in FVC in L
Description: Decline (change) in FVC is presented from Week 0 to Week 12. FVC was assessed using standardized spirometry equipment.
Time Frame: Week 0/Visit 2 up to Week 12
Population: Intent-to-treat Population: The ITT population included any randomized participants. The ITT Population was used for summary of demographic and baseline characteristics, and it was used for analysis of secondary endpoints except PK analysis
Measure: Mean (Standard Deviation); unit: L
Arm/Group | INS018_055 30 mg QD | INS018_055 30 mg BID | INS018_055 60 mg QD | Placebo
Number analyzed (Participants) | 13 | 12 | 10 | 14
L | -0.0270 (0.11368) | 0.0197 (0.14177) | 0.0984 (0.14113) | -0.0203 (0.18300)
Statistical Analysis 1: Comparison: INS018_055 30 mg QD; Test type: Other; Least Squares Mean = -0.0242, 95% CI 2-sided [-0.1050 to 0.0566], Standard Error of Mean 0.04121
Statistical Analysis 2: Comparison: INS018_055 30 mg BID; Test type: Other; Least Squares Mean = 0.0194, 95% CI 2-sided [-0.0687 to 0.1074], Standard Error of Mean 0.04492
Statistical Analysis 3: Comparison: INS018_055 60 mg QD; Test type: Other; Least Squares Mean = 0.0892, 95% CI 2-sided [-0.0087 to 0.1872], Standard Error of Mean 0.04994
Statistical Analysis 4: Comparison: Placebo; Test type: Other; Least Squares Mean = -0.0082, 95% CI 2-sided [-0.0981 to 0.0817], Standard Error of Mean 0.04585

4. Secondary Outcome: Absolute Change in FVC % Predicted
Description: Absolute change in FVC % predicted from Week 0 to Week 12 is presented. FVC was assessed using standardized spirometry equipment
Time Frame: Week 0/Visit 2 up to Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent predicted
Arm/Group | INS018_055 30 mg QD | INS018_055 30 mg BID | INS018_055 60 mg QD | Placebo
Number analyzed (Participants) | 13 | 12 | 10 | 14
Percent predicted | -0.6729 (2.92554) | 0.6455 (3.73482) | 3.0461 (4.38853) | -0.5675 (5.44712)
Statistical Analysis 1: Comparison: INS018_055 30 mg QD; Test type: Other; Least Squares Mean = -0.6043, 95% CI 2-sided [-2.9549 to 1.7462], Standard Error of Mean 1.19916
Statistical Analysis 2: Comparison: INS018_055 30 mg BID; Test type: Other; Least Squares Mean = 0.6510, 95% CI 2-sided [-1.9603 to 3.2624], Standard Error of Mean 1.33193
Statistical Analysis 3: Comparison: INS018_055 60 mg QD; Test type: Other; Least Squares Mean = 2.4975, 95% CI 2-sided [-0.3187 to 5.3136], Standard Error of Mean 1.43617
Statistical Analysis 4: Comparison: Placebo; Test type: Other; Least Squares Mean = -0.0209, 95% CI 2-sided [-2.8142 to 2.7724], Standard Error of Mean 1.42470

5. Secondary Outcome: Relative Change in FVC % Predicted
Description: Relative change in FVC % predicted from Week 0 to Week 12 is presented. FVC was assessed using standardized spirometry equipment
Time Frame: Week 0/Visit 2 up to Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent predicted
Groups:
- INS018_055 60 mg QD: Group 3: INS018_055 once daily up to 12 weeks, high dose INS018_055: Pharmaceutical formulation: Capsules Mode of administration:Oral
Arm/Group | INS018_055 30 mg QD | INS018_055 30 mg BID | INS018_055 60 mg QD | Placebo
Number analyzed (Participants) | 13 | 12 | 10 | 14
Percent predicted | -0.6724 (4.05537) | 0.4434 (5.96895) | 3.2194 (5.28129) | -0.8414 (8.31651)
Statistical Analysis 1: Comparison: INS018_055 30 mg QD; Test type: Other; Least Squares Mean = -0.5762, 95% CI 2-sided [-4.0035 to 2.8511], Standard Error of Mean 1.74854
Statistical Analysis 2: Comparison: INS018_055 30 mg BID; Test type: Other; Least Squares Mean = 0.5884, 95% CI 2-sided [-3.1449 to 4.3216], Standard Error of Mean 1.90433
Statistical Analysis 3: Comparison: INS018_055 60 mg QD; Test type: Other; Least Squares Mean = 2.6554, 95% CI 2-sided [-1.8486 to 7.1593], Standard Error of Mean 2.29650
Statistical Analysis 4: Comparison: Placebo; Test type: Other; Least Squares Mean = -0.0625, 95% CI 2-sided [-4.3227 to 4.1977], Standard Error of Mean 2.17274

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from the signing of the informed consent form (ICF) until end of study (EOS) visit i.e. up to 13 weeks (+10 days).
Description: An AE is any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with a medicinal product, whether or not related. The following are also recorded as an AE: worsening of pre-existing conditions and clinically relevant changes in tests (as per the investigator).
  Within a system organ class and preferred term, participants may report >1 AE. Participants are counted once per relationship, preferred term, and system organ class.
Arm/Group | INS018_055 30 mg QD | INS018_055 30 mg BID | INS018_055 60 mg QD | Placebo
All-Cause Mortality (participants affected / at risk) | 0/18 | 1/18 | 0/18 | 0/17
Serious Adverse Events (participants affected / at risk) | 2/18 | 4/18 | 7/18 | 3/17
Other Adverse Events (participants affected / at risk) | 13/18 | 15/18 | 15/18 | 12/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | INS018_055 30 mg QD (N=18) | INS018_055 30 mg BID (N=18) | INS018_055 60 mg QD (N=18) | Placebo (N=17)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Liver injury (Hepatobiliary disorders) | 0 | 1 | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 2 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 1 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0 | 0
Chronic gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Chest discomfort (General disorders) | 0 | 0 | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | INS018_055 30 mg QD (N=18) | INS018_055 30 mg BID (N=18) | INS018_055 60 mg QD (N=18) | Placebo (N=17)
Alanine aminotransferase increased (Investigations) | 1 | 1 | 6 | 1
Blood bilirubin increased (Investigations) | 0 | 1 | 4 | 2
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 2 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 2 | 0
Blood urea increased (Investigations) | 0 | 1 | 1 | 0
C-reactive protein increased (Investigations) | 1 | 1 | 0 | 0
Carbohydrate antigen 19-9 increased (Investigations) | 0 | 1 | 1 | 0
Protein urine present (Investigations) | 1 | 1 | 0 | 0
Red blood cell sedimentation rate increased (Investigations) | 0 | 1 | 1 | 0
Weight decreased (Investigations) | 0 | 1 | 0 | 1
Alpha hydroxybutyrate dehydrogenase increased (Investigations) | 0 | 0 | 1 | 0
Bile acids increased (Investigations) | 0 | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 1
Blood creatine phosphokinase MB increased (Investigations) | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0
Blood fibrinogen increased (Investigations) | 1 | 0 | 0 | 0
Blood glucose increased (Investigations) | 0 | 0 | 1 | 0
Blood pressure increased (Investigations) | 0 | 0 | 1 | 0
Carbon dioxide decreased (Investigations) | 0 | 1 | 0 | 0
Carotid intima-media thickness increased (Investigations) | 1 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 0 | 0
Electrocardiogram ST segment abnormal (Investigations) | 1 | 0 | 0 | 0
Electrocardiogram T wave abnormal (Investigations) | 0 | 1 | 0 | 0
Electrocardiogram high voltage (Investigations) | 0 | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 0
Glutamate dehydrogenase increased (Investigations) | 0 | 1 | 0 | 0
Hepatic enzyme abnormal (Investigations) | 0 | 0 | 1 | 0
Immunoglobulins increased (Investigations) | 0 | 0 | 1 | 0
Interferon gamma level increased (Investigations) | 0 | 0 | 1 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 1 | 0
Low density lipoprotein increased (Investigations) | 0 | 0 | 1 | 0
Neutrophil count increased (Investigations) | 1 | 0 | 0 | 0
QRS axis abnormal (Investigations) | 1 | 0 | 0 | 0
Red blood cells urine positive (Investigations) | 0 | 0 | 1 | 0
Reticulocyte count increased (Investigations) | 0 | 0 | 1 | 0
Throxine free decreased (Investigations) | 0 | 1 | 0 | 0
Tri-iodothyronine increased (Investigations) | 1 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 1 | 0
White blood cell count increased (Investigations) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 4 | 1 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1 | 2 | 3
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 2
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 1 | 0 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 1 | 0
Soft tissue infection (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 3 | 5 | 4 | 2
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 2 | 1 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 1 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Hyperchloraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 2 | 4 | 3 | 2
Liver injury (Hepatobiliary disorders) | 0 | 2 | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 2 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hepatic steatosis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 3 | 5 | 0
Abdominal discomfort (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 1
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Eosinophilia myalgia syndrome (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Atrioventricular block first degree (Cardiac disorders) | 1 | 0 | 1 | 0
Supraventricular extrasystoles (Cardiac disorders) | 2 | 0 | 0 | 0
Aortic valve incompetence (Cardiac disorders) | 1 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1
Bundle branch block left (Cardiac disorders) | 1 | 0 | 0 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 0 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 1 | 0
Eye swelling (Eye disorders) | 1 | 0 | 0 | 0
Periorbital oedema (Eye disorders) | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0
Xerophthalmia (Eye disorders) | 0 | 0 | 1 | 0
Chest discomfort (General disorders) | 0 | 0 | 1 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 2 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Prostatic calcification (Reproductive system and breast disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2024-02-02): https://cdn.clinicaltrials.gov/large-docs/20/NCT05938920/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-06): https://cdn.clinicaltrials.gov/large-docs/20/NCT05938920/SAP_001.pdf